CLINICAL TRIAL: NCT00513331
Title: The Valley Hospital Center for Barrett's Esophagus and Gastroesophageal Reflux Disease (GERD)
Brief Title: Barrett's Esophagus & Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: Valley Health System (Other)
Responsible Party: Sponsor
Other Study IDs: VHS07.0017
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Barrett's Esophagus; GERD
Keywords: Barrett's Esophagus; GERD; Carcinoma
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux; Carcinoma | interventions — Endoscopy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood for future analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Algorithm #1: Patients without visable lesions
  Interventions: Procedure: Endoscopy
- Algorithm #2: Patients with a visable lesion that is less than 1cm
  Interventions: Procedure: Endoscopy; Procedure: Radiofrequency ablation protocol; Procedure: Endoscopic mucosal resection protocol
- Algorithm #3: Patients with a visable lesion greater than 1cm
  Interventions: Procedure: Endoscopy; Procedure: Radiofrequency ablation protocol; Procedure: Endoscopic mucosal resection protocol

INTERVENTIONS:
Procedure: Endoscopy — Initial Assessment for lesions can be based on information obtained from previous upper endoscopies and or pathology reports. Repeat Endoscopic assessments are based on initial and follow-up assessments.
Procedure: Radiofrequency ablation protocol — Ablation using the HALO 360 system according to protocol established by BARRX, Inc.
  Groups: Algorithm #2; Algorithm #3
Procedure: Endoscopic mucosal resection protocol — Excision of lesion using DUETTE, marketed by Wilson-Cook
  Groups: Algorithm #2; Algorithm #3

SUMMARY:
This is a study of Barrett's Esophagus (BE) and Gastroesophageal Reflux Disease (GERD). It aims to look at the long term efficacy of evidence-based cutting edge diagnostic and therapeutic algorithms and techniques such as radiofrequency ablation, endoscopic mucosal resection and surveillance endoscopy with biopsy. Additionally, biological analyses will be performed in hopes of identifying biomarkers associated with the progression of BE to esophageal cancer.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a known premalignant condition of the esophagus, predisposing to the development of esophageal adenocarcinoma. BE represents a change in the lining (mucosa) of the esophagus which is known to be produced as a result of chronic gastroesophageal reflux. The current standard of care for patients with BE includes serial performance of upper endoscopy with multiple biopsies, performed at designated time intervals. However, the emergence of new technologies for the management of this condition has made the care of these patients non-uniform, and subject to biases of individual treating physicians.

The protocol at The Valley Hospital and Blumenthal Cancer Center aims to standardize the management of patients with Barrett's esophagus, with and without dysplasia, using evidence-based, cutting edge diagnostic and therapeutic algorithms and techniques such as radiofrequency ablation, endoscopic mucosal resection, and surveillance endoscopy with biopsies. If biopsies suggest the development of carcinoma or high grade dysplasia surgical removal of the esophagus is recommended. This study aims to look at the long-term efficacy of these procedures. In addition, data regarding clinical outcomes will be collected as well as blood, tissue and surgical specimens for proteomic analysis in hopes of identifying biomarkers associated with the progression of dysplasia to adenocarcinoma. Although patients will ultimately make their own informed decisions regarding the management of their BE, this protocol serves to unify physician recommendations, and allows for the collection and interpretation of data.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 85.
* Patient must have Barrett's Esophagus. Patients may be enrolled based on previous endoscopy reports and/or pathology reports. It is not necessary that each patient have endoscopy for the sole purpose of enrollment.
* Must agree to allow their clinical information to be collected, stored, analyzed and reported.
* Must allow portions of their biopsy/surgical specimens to be collected, stored, analyzed and reported.
* Must agree to fill out patient questionnaires in conjunction with the research study assistant assigned to this protocol (either in person or via telephone contact) at designated timepoints.

Exclusion Criteria:

* Intestinal metaplasia of the cardia, without an esophageal columnar lining.
* Unable to provide informed consent.
* Unable or unwilling to undergo endoscopic procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Referred Patients with underlying disease of BE or GERD
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2007-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To standardize physician recommendations and provide cutting edge technology to patients with BE and GERD, and establish a Valley Hospital Center for Barrett's Esophagus and GERD | Until study complete

SECONDARY OUTCOMES:
To collect and store patient data regarding their Barrett's esophagus | Througout Study
To collect tissue specimens (biopsy and surgical specimens) for use in proteomic analysis to investigate the dysplasia/carcinoma sequence at the protein expression level. | throughout Study
To assess clinical outcomes of patients enrolled in The Valley Hospital Center for Barrett's Esophagus and GERD, and modify algorithms as appropriate. | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Korst, MD, Principal Investigator — Valley Health Systems/ The Valley Hospital
Locations (1):
- Valley Health System - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey, United States